CLINICAL TRIAL: NCT04381026
Title: Study on the Effect of a Nutritional Supplement With Isoflavones on the Symptoms of Climacteric in Healthy Women
Brief Title: Effects of a New Botanical Extracts Combination on Quality of Life in Menopausal Spanish Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nektium Pharma SL (Industry)
Collaborators: Clínica Barem (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO_WH_HCT_2016.01
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Menopause; Dietary Supplements; Quality of Life
Keywords: Menopause; Hot flushes; Isoflavones; Aframomum melegueta extract; Punica granatum extract; Cervantes Scale
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Pill of 500 mg containing filler agent, two pills daily for eight weeks.
  Interventions: Dietary Supplement: Placebo
- Treatment Group with botanical extracts (Experimental): Pill of 500 mg containing botanicals and filler agent, two pills daily for eight weeks.
  Interventions: Dietary Supplement: Botanical dry extracts combination

INTERVENTIONS:
Dietary Supplement: Botanical dry extracts combination — Aframomum melgueta dry extract (50mg), Glycine max bean dry extract (100mg) and Punica granatum skin extract (100mg)
  Arms: Treatment Group with botanical extracts
Dietary Supplement: Placebo — Filler agent
  Arms: Placebo Group

SUMMARY:
This study was designed to evaluate the beneficial effects and safety of a standardised botanical extract combination containing soy isoflavone extract, grains of paradise seed dry extract and pomegranate skin dry extract on health-related Quality of Life in healthy Spanish menopausal women with hot flashes, anxiety, and depressive symptoms using the self reported and validated Cervantes Scale.

DETAILED DESCRIPTION:
Fifty-seven outpatient women (45-65 years) with menstrual problems associated with climacteric syndrome were enrolled from April 2018 to April 2019 in the context of a prospective, placebo-controlled, double-blind study. Women were randomized to receive treatment with either the botanical combination (250 mg daily divided into two doses) or placebo for eight weeks. At the beginning and end of the study, health-related Quality of Life was assessed using the Cervantes Scale.

ELIGIBILITY:
Inclusion Criteria:

* Women in the Climacteric Phase under medical criteria based on Health questionnaire, Blood and urine test.
* Informed consent to participate in the study.

Exclusion Criteria:

* Hormone-related pathologies.
* Menopause from surgery origin.
* Family or personal history of endocrine cancer.
* Known hypersensitivity to gluten, soybeans, soy protein, dairy products, pomegranate or grains of paradise.
* Vegetarian diet or daily consumption of soya rich-products during the last year.
* Anovulatory treatment.
* Hormone replacement treatment.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 8 in the global score of quality of life using the validated Cervantes Scale | 8 weeks
  To evaluate the improvement of quality of life after trial, a variable to quantify the percentage of reduction between after-treatment and before-treatment for global score (GS) in quality of life is generated: [Variation%=100 x ((initial GS value-final GS value)/ initial GS value)]

SECONDARY OUTCOMES:
Change from Baseline to Week 8 in the Menopause-health score of quality of life using the validated Cervantes Scale | 8 weeks
  To evaluate the improvement of quality of life after trial, a variable to quantify the percentage of reduction between after-treatment and before-treatment for Menopause and health score (MHS) in quality of life is generated: [Variation%=100 x ((initial MHS value-final MHS value)/ initial MHS value)]
Change from Baseline to Week 8 in the psychic score of quality of life using the validated Cervantes Scale | 8 weeks
  To evaluate the improvement of quality of life after trial, a variable to quantify the percentage of reduction between after-treatment and before-treatment for psychic score (PS) in quality of life is generated: [Variation%=100 x ((initial PS value-final PS value)/ initial PS value)]
Change from Baseline to Week 8 in the sexuality-couple score of quality of life using the validated Cervantes Scale. | 8 weeks
  To evaluate the improvement of quality of life after trial, a variable to quantify the percentage of reduction between after-treatment and before-treatment for sexuality-couple score (SCS) in quality of life is generated: [Variation%=100 x ((initial SCS value-final SCS value)/ initial SCS value)]

OTHER OUTCOMES:
Change from baseline to week 8 in the bogy weight | 8 weeks
  To evaluate the body weight reduccion, a variable to quantify the percentage of reduction between after-treatment and before-treatment in body weight (BW) is generated: [Variation%=100 x ((initial BW value-final BW value)/ initial BW value)]

CONTACTS AND LOCATIONS:
Overall Officials: Laura López-Ríos, PhD, Principal Investigator — Nektium Pharma SL
Locations (1):
- Clinica Barem, Las Palmas de Gran Canaria, Las Palmas (Canary Islands), Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greene JG. Constructing a standard climacteric scale. Maturitas. 1998 May 20;29(1):25-31. doi: 10.1016/s0378-5122(98)00025-5. PMID 9643514
- [Result] Buendia Bermejo J, Rodriguez Segarra R, Yubero Bascunana N, Martinez Vizcaino V. [Design and validation of a questionnaire in Spanish for measuring the quality of life in postmenopausal women: the MENCAV questionnaire]. Aten Primaria. 2001 Feb 15;27(2):94-100. doi: 10.1016/s0212-6567(01)78780-x. Spanish. PMID 11256098
- [Result] Palacios S, Ferrer-Barriendos J, Parrilla JJ, Castelo-Branco C, Manubens M, Alberich X, Marti A; Grupo Cervantes. [Health-related quality of life in the Spanish women through and beyond menopause. Development and validation of the Cervantes Scale]. Med Clin (Barc). 2004 Feb 21;122(6):205-11. doi: 10.1016/s0025-7753(04)74198-6. Spanish. PMID 15012887
- [Result] Heinemann K, Ruebig A, Potthoff P, Schneider HP, Strelow F, Heinemann LA, Do MT. The Menopause Rating Scale (MRS) scale: a methodological review. Health Qual Life Outcomes. 2004 Sep 2;2:45. doi: 10.1186/1477-7525-2-45. PMID 15345062
- [Result] Low Dog T. Menopause: a review of botanical dietary supplements. Am J Med. 2005 Dec 19;118 Suppl 12B:98-108. doi: 10.1016/j.amjmed.2005.09.044. PMID 16414334
- [Result] Tranche S, Brotons C, Pascual de la Pisa B, Macias R, Hevia E, Marzo-Castillejo M. Impact of a soy drink on climacteric symptoms: an open-label, crossover, randomized clinical trial. Gynecol Endocrinol. 2016 Jun;32(6):477-82. doi: 10.3109/09513590.2015.1132305. Epub 2016 Jan 25. PMID 26806546
- [Result] Kang SJ, Choi BR, Kim SH, Yi HY, Park HR, Kim DC, Choi SH, Han CH, Park SJ, Song CH, Ku SK, Lee YJ. Dried pomegranate potentiates anti-osteoporotic and anti-obesity activities of red clover dry extracts in ovariectomized rats. Nutrients. 2015 Apr 9;7(4):2622-47. doi: 10.3390/nu7042622. PMID 25912038
- [Result] Balk E, Chung M, Chew P, Ip S, Raman G, Kupelnick B, Tatsioni A, Sun Y, Wolk B, DeVine D, Lau J. Effects of soy on health outcomes. Evid Rep Technol Assess (Summ). 2005 Aug;(126):1-8. doi: 10.1037/e439502005-001. No abstract available. PMID 16194125
- [Result] Ferrari A. Soy extract phytoestrogens with high dose of isoflavones for menopausal symptoms. J Obstet Gynaecol Res. 2009 Dec;35(6):1083-90. doi: 10.1111/j.1447-0756.2009.01058.x. PMID 20025635
- [Result] Klein MA, Nahin RL, Messina MJ, Rader JI, Thompson LU, Badger TM, Dwyer JT, Kim YS, Pontzer CH, Starke-Reed PE, Weaver CM. Guidance from an NIH workshop on designing, implementing, and reporting clinical studies of soy interventions. J Nutr. 2010 Jun;140(6):1192S-1204S. doi: 10.3945/jn.110.121830. Epub 2010 Apr 14. PMID 20392880
- [Result] Munro IC, Harwood M, Hlywka JJ, Stephen AM, Doull J, Flamm WG, Adlercreutz H. Soy isoflavones: a safety review. Nutr Rev. 2003 Jan;61(1):1-33. doi: 10.1301/nr.2003.janr.1-33. PMID 12638461
- [Result] Satpathy S, Patra A, Purohit AP. Estrogenic activity of Punica granatum L. peel extract. Asian Pacific J. Reprod. 2013; 2(1): 19-24
- [Result] Bialonska D, Ramnani P, Kasimsetty SG, Muntha KR, Gibson GR, Ferreira D. The influence of pomegranate by-product and punicalagins on selected groups of human intestinal microbiota. Int J Food Microbiol. 2010 Jun 15;140(2-3):175-82. doi: 10.1016/j.ijfoodmicro.2010.03.038. Epub 2010 Apr 2. PMID 20452076
- [Result] Mori-Okamoto J, Otawara-Hamamoto Y, Yamato H, Yoshimura H. Pomegranate extract improves a depressive state and bone properties in menopausal syndrome model ovariectomized mice. J Ethnopharmacol. 2004 May;92(1):93-101. doi: 10.1016/j.jep.2004.02.006. PMID 15099854
- [Result] Ilic NM, Dey M, Poulev AA, Logendra S, Kuhn PE, Raskin I. Anti-inflammatory activity of grains of paradise (Aframomum melegueta Schum) extract. J Agric Food Chem. 2014 Oct 29;62(43):10452-7. doi: 10.1021/jf5026086. Epub 2014 Oct 20. PMID 25293633
- [Result] Sugita J, Yoneshiro T, Hatano T, Aita S, Ikemoto T, Uchiwa H, Iwanaga T, Kameya T, Kawai Y, Saito M. Grains of paradise (Aframomum melegueta) extract activates brown adipose tissue and increases whole-body energy expenditure in men. Br J Nutr. 2013 Aug;110(4):733-8. doi: 10.1017/S0007114512005715. Epub 2013 Jan 11. PMID 23308394
- [Result] Igwe SA, Emeruwa IC, Modie JA. Ocular toxicity of Afromomum melegueta (alligator pepper) on healthy Igbos of Nigeria. J Ethnopharmacol. 1999 Jun;65(3):203-6. doi: 10.1016/s0378-8741(98)00188-3. PMID 10404417
- [Derived] Lopez-Rios L, Barber MA, Wiebe J, Machin RP, Vega-Morales T, Chirino R. Influence of a new botanical combination on quality of life in menopausal Spanish women: Results of a randomized, placebo-controlled pilot study. PLoS One. 2021 Jul 21;16(7):e0255015. doi: 10.1371/journal.pone.0255015. eCollection 2021. PMID 34288973
- See also: Clinical guides for menopause from AEEM — https://aeem.es/para-profesionales/guias-clinicas/
- See also: paper on Validity and reliability of the Kupperman test [Spanish] — https://www.elsevier.es/es-revista-clinica-e-investigacion-ginecologia-obstetricia-7-articulo-validez-fiabilidad-prueba-kupperman-S0210573X08730612